CLINICAL TRIAL: NCT06596954
Title: Lymphocyte-sparing Thoracic Radiotherapy vs Conventional Radiotherapy for Esophageal Squamous Cell Carcinoma Treated With Neoadjuvant Therapy: an Open Label, Randomized Controlled Trial
Brief Title: Lymphocyte-sparing Thoracic Radiotherapy for Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, QIWEIXIANG, Deputy Chief Physician, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-210
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2024-09

CONDITIONS: Esophageal Squamous Cell Cancer
Keywords: esophageal cancer; neoadjuvant treatment; lymphocyte-sparing radiotherapy; prognosis
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lymphocyte-sparing radiotherapy (Experimental): Firstly, ensure coverage of the PTV (Planning Target Volume). Secondly, limit the doses to the heart, bilateral lungs, and spinal cord to meet the required dose constraints. While maintaining target coverage and traditional OAR (Organs At Risk) dose constraints, also address dose limits for the TVB1-12 thoracic vertebral bodies, ribs, spleen, and major thoracic blood vessels to protect the lymphocyte
- conventional radiotherapy (Active Comparator): ensure coverage of the PTV (Planning Target Volume) and limit the doses to the heart, bilateral lungs, and spinal cord to meet the required dose constraints. do not limits the dose for lymphocyte-related organs

INTERVENTIONS:
Radiation: lymphocyte-sparing radiotherapy — the radiotherapy regimen is 41.4Gy/23Fx. Ensure 95% coverage of the PTV (Planning Target Volume) and limit the doses to the heart, bilateral lungs, and spinal cord to meet the required dose constraints. While maintaining target coverage and traditional OAR (Organs At Risk) dose constraints, also address dose for lymphocyte-relate organs including the TVB1-12 thoracic vertebral bodies, ribs, spleen, and major thoracic blood vessels.
Radiation: conventional radiotherapy — the radiotherapy regimen is 41.4Gy/23Fx. Ensure 95% coverage of the PTV (Planning Target Volume) and limit the doses to the heart, bilateral lungs, and spinal cord to meet the required dose constraints. do not limit dose for lymphocyte-relate organs including the TVB1-12 thoracic vertebral bodies, ribs, spleen, and major thoracic blood vessels.

SUMMARY:
Esophageal squamous cell carcinoma (ESCC) is one of the most aggressive malignant tumors. Although neoadjuvant chemoradiotherapy combined with surgery has significantly improved the survival rate of patients with locally advanced esophageal cancer, approximately half of the patients will experience local regional recurrence or distant metastasis. Lymphocytes are crucial immune cells in the human body, playing a key role in combating infections and tumor development. In recent years, an increasing body of research has indicated that lymphocyte depletion is a significant factor associated with poor prognosis in various solid tumors, including esophageal cancer. The lymphocyte depletion caused by radiotherapy has garnered considerable attention from oncologists. However, there is still a lack of prospective clinical research data on lymphocyte protection in thoracic tumors. Therefore, this study aims to provide high-level evidence from evidence-based medicine regarding the correlation between lymphocyte depletion and prognosis in esophageal cancer patients, offering more effective strategies and methods to improve the outcomes of neoadjuvant chemoradiotherapy for esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are able to understand and are willing to participate in the trial, and a signed consent form can be obtained;
2. Pathologically confirmed esophageal squamous cell carcinoma;
3. locally advanced ESCC (cT3-4 or N+);
4. the age of patients should be more than 18 years, and less than 80 years;
5. aged between 18 and 80 years;
6. KPS score of patients should be more than 80

Exclusion Criteria:

1. diagnosis of metastatic esophageal cancer;
2. Patient refuses to receive systemic drug treatment;
3. clinical diagnosis of pleural metastasis or malignant pleural effusion;
4. Pregnant or breastfeeding women;
5. Severe non-cancerous medical comorbidities that affect the implementation of radiotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
acute grade 3/4 lymphopenia | 1 months after surgery
  from treatment to 1 months after completion of neoadjuvant chemoradiotherapy

SECONDARY OUTCOMES:
Lymphocyte-sparing radiotherapy plan pass rate in lymphocyte-sparing group | within 1 week after completion of neoadjuvat radiotherapy plan;
  the pass rate of the esophageal cancer lymphocyte-sparing plan is evaluated without compromising target volume coverage and conventional normal tissue constraints (heart, lungs, and spinal cord)
Incidence of grade 3 or higher hematologic toxicity | from neoadjuvant chemoradiotherapy to 1 monther after completion of neoadjuvant chemoradiotherapy
  The incidence of grade 3 or higher hematologic toxicity during nCRT and within 1 month after treatment between lymphocyte-sparing RT group and conventional RT group.
Pathological complete response rate (pCR) | 1 months after surgery
  The pCR rate in ESCC patients who underwent nCRT and radical surgery between lymphocyte-sparing RT group and conventional RT group.
R0 resection rate | 1 month after surgery
  the R0 resection rate in ESCC patients who underwent nCRT and radical surgery between lymphocyte-sparing RT group and conventional RT group.
Postoperative complications | 1 month after surgery
  which was defined as 30-day postoperative complications graded according to the Clavien-Dindo classification;
recurrence-free survival | 2 year
  from completion of surgery to any recurrence
Overall survival | 3 years
  from treatment to death

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital, Shanghai jiaotong university school of medicine, Shanghai, China, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qi WX, Li S, Li H, Zhang S, Cai G, Xu C, Zhang Y, Chen J, Zhao S. Sparing lymphocytes during preoperative adjuvant radiotherapy for oesophageal squamous cell carcinoma (SPARE): protocol for an open-label, randomised controlled trial. BMJ Open. 2025 Sep 21;15(9):e096803. doi: 10.1136/bmjopen-2024-096803. PMID 40976677